CLINICAL TRIAL: NCT06824948
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Multiple-Dose Phase I Clinical Study to Evaluate the Safety, Tolerance, and Pharmacokinetic Profiles of Timolol Maleate Gel in Healthy Chinese Adult Subjects
Brief Title: Evaluate the Safety, Tolerance, and Pharmacokinetic Profiles of Timolol Maleate Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Auson Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASN001C001; CRC-C1824 (Other: China Drug Trials)
Record Dates: First submitted 2025-01-23; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 2-0.5%TM (Experimental): Participants will be randomized to receive 0.5%TM or matching placebo 2 times a day.
  Interventions: Drug: Timolol Maleate Gel; Drug: Placebo
- Group 3-0.5%TM (Experimental): Participants will be randomized to receive 0.5%TM or matching placebo 3 times a day.
  Interventions: Drug: Timolol Maleate Gel; Drug: Placebo
- Group 1-0.5%TM (Experimental): Participants will be randomized to receive 0.5%TM or matching placebo 1 time a day.
  Interventions: Drug: Timolol Maleate Gel; Drug: Placebo

INTERVENTIONS:
Drug: Timolol Maleate Gel — A 2-day washout phase follows 1 dose on Day 1, the subjects are applied with 0.5% timolol maleate gel one time a day during Day 3-Day 12.
  Arms: Group 1-0.5%TM
Drug: Placebo — A 2-day washout phase follows 1 dose on Day 1, the subjects are applied with placebo one time a day during Day 3-Day 12.
  Arms: Group 1-0.5%TM
Drug: Timolol Maleate Gel — A 2-day washout phase follows 1 dose on Day 1, the subjects are applied with 0.5% timolol maleate gel 2 times a day during Day 3-Day 12.
  Arms: Group 2-0.5%TM
Drug: Placebo — A 2-day washout phase follows 1 dose on Day 1, the subjects are applied with placebo 2 times a day during Day 3-Day 12.
  Arms: Group 2-0.5%TM
Drug: Timolol Maleate Gel — A 2-day washout phase follows 1 dose on Day 1, the subjects are applied with 0.5% timolol maleate gel 3 times a day during Day 3-Day 12.
  Arms: Group 3-0.5%TM
Drug: Placebo — A 2-day washout phase follows 1 dose on Day 1, the subjects are applied with placebo 3 times a day during Day 3-Day 12.
  Arms: Group 3-0.5%TM

SUMMARY:
The goal of this clinical trial is to to evaluate the safety, tolerance, and pharmacokinetic profiles of Timolol Maleate Gel in healthy Chinese adult subjects. The main questions aim to answer are:

• The pharmacokinetic endpoints: Single dose:Tmax, Cmax, etc. Multiple doses:AUC0-t, AUC0-inf, λz, t1/2, etc.

• The safety and tolerance endpoints: Physical examination, vital signs, 12-lead ECG, laboratory tests (hematology, blood biochemistry and urinalysis), adverse events, local tolerance.

Researchers will compare TM gel to a placebo (a look-alike substance that contains no drug) to see if TM gel works to treat IH.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female subjects aged 18-55 years (including the cut point, subject to the time of signing the ICF);
2. Subjects with the body mass index (BMI) of 19-26 kg/m2 (including the cut point), where the body weight should be ≥ 50 kg for male subjects and ≥ 45 kg for female subjects;
3. Subjects who have no pregnancy plan, voluntarily adopt effective birth controls, and have no sperm donation or egg donation plan during the study until 3 months after the last dose. For specific birth controls, see Appendix 1: Birth Control, Definition of Female Subjects of Childbearing Age, and Contraception Requirements;
4. Subjects fully understand the study objective, nature, methods and possible adverse reactions, voluntarily become subjects, and sign the ICFs;
5. Subjects who have no skin damage or scar or skin disease at the administration site; Subjects who can complete the trial as required in the protocol.

Exclusion Criteria:

1. Subjects who are allergic to timolol maleate and similar drugs;
2. Subjects who have any difficulty in venous blood collection;
3. Subjects who have cardiogenic shock, Grade I or Grade III atrioventricular block, cardiac failure, sinus bradycardia, hypotension, and CS as assessed by the study physician;
4. Subjects who have bronchial asthma, airway sensitive disease, ventilation difficult or other pulmonary disorders;
5. Subjects who have had a history of drug abuse in the past five years or used drugs within the 3 months before the study; or subjects who are positive in the drug abuse screening test in the screening phase;
6. Subjects who have smoked more than 5 cigarettes a day within the 3 months before screening;
7. Subjects who have consumed more than 14 units of alcohol (1 unit of alcohol = 360 mL beer or 45 mL 40% spirits or 150 mL wine) weekly within 6 months before the screening or have taken alcohol-containing products 48 h pre-dose, or were or positive in the alcohol breath test in the screening phase and/or the baseline phase;
8. Subjects who have used any drug that induces or inhibits liver metabolic enzymes within 28 days pre-dose in the study;
9. Subjects who have used any Rx, OTC or Chinese herbal medicine within 14 days pre-dose in the study;
10. Subjects who have took food or drink (such as grapefruit) containing enzymes that can induce or inhibit liver metabolism within 7 days pre-dose in the study;
11. Subjects who have ingested any food or drink containing caffeine or xanthine (e.g., coffee, tea, chocolate) during the period at 48 ho pre-dose to completion of the last PK blood sampling;
12. Subjects who have diseases or factors with clinical abnormalities, including but not limited to neurological, cardiovascular, blood, liver, kidney, gastrointestinal, respiratory, metabolic, endocrine, immune, skeletal system diseases or other factors;
13. Results of the vital signs assessment, physical examinations, laboratory test, 12-lead electrocardiogram and chest radiograph showed CS;
14. Subjects who are human immunodeficiency virus (HIV) antibody positive, hepatitis B surface antigen positive, hepatitis C virus antibody positive, or syphilis antibody positive;
15. Female subjects who are positive for pregnancy test in the screening phase or the baseline phase or who are breastfeeding;
16. Subjects who have had a clinically significant major disease or major surgical procedure within 4 weeks prior to dosing, or was expected to require major surgery during the study;
17. Subjects who have participated in other clinical drug trials within 3 months pre-dose in the study;
18. Subjects who have donated blood or blood loss > 400 mL within 3 months before screening; Any other circumstances that may affect the subjects in providing ICFs or following the study protocol, or participation in the study may affect the study results or the subjects' own safety as assessed by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Local tolerance | 13 Days
  Local tolerance will be evaluated by an investigator or designated evaluator (e.g., dermatologist) using the blinding method.The intensity (e.g., No evidence of irritation;Minimal erythema that is barely perceptible;Definite erythema that is readily visible and minimal edema or minimal papular response;Erythema and papules, et al) of the skin response is assessed on a 8 point scale.Other response score is assessed from "A" to "H".
Adverse events | Throughout study completion, an average 13 days
  Frequency, severity and relatedness of adverse events
Vital signs (blood pressure) | the screening phase, Day -1, Day 1, 3, 6, 9, 12, and Day 13.
  Number of participants with clinically significant changes in vital signs (blood pressure)
Vital signs (temperature) | the screening phase, Day -1, Day 1, 3, 6, 9, 12, and Day 13.
  Number of participants with clinically significant changes in vital signs (temperature)
Vital signs (pulse rate) | the screening phase, Day -1, Day 1, 3, 6, 9, 12, and Day 13.
  Number of participants with clinically significant changes in vital signs (pulse rate)
Laboratory tests | the screening phase, the baseline phase, and on Days 6 and 13.
  Number of participants with clinical laboratory abnormalities (including hematology, blood biochemistry and urinalysis).
Physical examinations | the screening phase, baseline phase and on Day 13
  Number of participants with clinically significant changes in physical examinations.
12-lead ECG | the screening phase, baseline phase, Day 1, 3, 6, 9, 12, and Day 13.
  Number of participants with clinically significant changes in 12-lead ECG.

SECONDARY OUTCOMES:
Tmax | Day1 to Day13
  The pharmacokinetics of single and multiple dose levels in participants will include peak time.
Cmax | Day1 to Day13
  The pharmacokinetics of single and multiple dose levels in participants will include peak concentration.
AUC0-t | Day1 to Day13
  The pharmacokinetics of single and multiple dose levels in participants will include area under drug concentration-time curve.
AUC0-inf | Day1 to Day13
  area under drug concentration-time curve (AUC0-t) from 0 to t for the last accurately measurable concentration, area under drug concentration-time curve from 0 to infinity
λz | Day1 to Day13
  The pharmacokinetics of single and multiple dose levels in participants will include elimination rate constant.
t1/2 | Day1 to Day13
  The pharmacokinetics of single and multiple dose levels in participants will include elimination half-life.
%AUCex | Day1 to Day13
  The pharmacokinetics of single and multiple dose levels in participants will include AUC extrapolation percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui District Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No